CLINICAL TRIAL: NCT03764410
Title: Evaluation of Periodontal Clinical Parameters and Blood Tests in Diabetic Patients Submitted to Non-surgical Periodontal Treatment
Brief Title: Evaluation of Non - Surgical Periodontal Therapy in Diabetic Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metropolitana de Santos (Other)
Responsible Party: Principal Investigator, CAIO VINICIUS G. ROMAN TORRES, Professor, Universidade Metropolitana de Santos
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SantosMU4
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Diabetes Mellitus, Type 2; Periodontal Diseases
Keywords: Diabetes mellitus, periodontal diseases, periodontal index
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Periodontal Diseases; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetic group DG (Experimental): Non-surgical periodontal treatment with scaling and root coronary planing, oral hygiene instructions and removal of biofilm retention factors
  Interventions: Procedure: Non-surgical periodontal treatment
- No diabetic group NG (Active Comparator): Non-surgical periodontal treatment with scaling and root coronary planing, oral hygiene instructions and removal of biofilm retention factors
  Interventions: Procedure: Non-surgical periodontal treatment

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — all the individuals included in the study received periodontal treatment with scaling and root planing with the use of local anesthesia and removal of factors that could cause biofilm retention such as fixed prosthesis, restorations, cervical abrasions. Four weekly sessions lasting 30 minutes each.

SUMMARY:
Unfavorable systemic conditions condition a low resistance of the host to the virulence of the aggressive agent, causing in a periodontal disease and may lead to difficulties in the therapeutic response. The longer the duration of diabetes, it is suggested that greater severity of periodontal disease and loss of insertion. The objective of the present study will be to evaluate the clinical, microbial and immunological characteristics in diabetic subjects with chronic periodontitis submitted to non-surgical periodontal treatment. Will be 120 individuals with chronic periodontitis, including 60 type 2 diabetic subjects and 60 healthy should receive and have access to the informed consent form. Medical and dental clinical examination should be performed and evaluation microbial and immunological properties of gingival fluid and saliva respectively. Non-surgical periodontal therapy with subgingival scaling should be performed in all individuals who will be evaluated at two times: at the beginning and after 90 days of the periodontal therapy with new performing clinical exams and collecting oral samples, oral hygiene instructions will be addressed in two sessions. The data will be subjected to appropriate statistical tests and shall provide a comparison between the times. There seems to be a relationship between type 2 diabetes and periodontal disease and studies that provide the implementation of therapy are essential for clarifying the relationship.

DETAILED DESCRIPTION:
There is a need for more intense metabolic control of the diabetic patient with periodontal disease, since the destruction of the periodontal tissues may be more aggressive, and a rapid control of the oral infection in these patients is essential to avoid the exacerbation of the metabolic imbalance. The initiation and progression of diabetes probably involve the interaction of a multiplicity of factors, these being hereditary and immunological factors that are governed by environmental factors. It can be observed that there is a lack of awareness of oral complications between diabetics and health care providers, and it is extremely important to understand how diabetes affects oral health and there is a need for regular follow-up of patients with diabetes mellitus by dentists and medical professional. The objective of the present study was to evaluate diabetic individuals with chronic periodontitis submitted to non-surgical periodontal treatment using clinical parameters and blood tests of fasting glycemia and glycated hemoglobin. The study was approved by the Research Committee of the Metropolitan University of Santos, nº 1.806.841 and all the patients involved in the research had access to the informed consent form. The diagnosis of diabetes was obtained through blood tests that test blood glucose levels, thus, before clinical evaluations, and 90 days after the periodontal treatment were performed fasting blood glucose tests. Healthy patients also underwent blood tests. After the anamnesis, periodontal clinical examination was performed by a previously trained and calibrated periodontist. Periodontal clinical parameters were realized. After periodontal therapy, all patients underwent further periodontal and laboratory blood tests. The data obtained were tabulated and received statistical treatment through the Anova and Chi square tests. There seems to be a relationship between type 2 diabetes and periodontal disease and studies that provide the implementation of therapy are essential for clarifying the relationship.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients with chronic periodontitis and Systemically healthy patients with chronic periodontitis

Exclusion Criteria:

* Patients who had any of the following characteristics were excluded from the study: use of orthodontic appliances, smoking, pregnancy or lactation, hepatitis or HIV infection or any other disease that compromises immune functions, immunosuppressive chemotherapy, antibiotics, phenytoin, calcium antagonists, cyclosporine or anti-inflammatory drugs one month before the initial consultation, use of oral contraceptives or hormone replacement, periodontal treatment in the 6 months prior to the start of the study.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2017-10-15 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
blood test fasting blood glucose | 90 days
  blood tests were performed at baseline and 90 days after periodontal therapy
blood test for glycated hemoglobin | 90 days
  blood tests were performed at baseline and 90 days after periodontal therapy

CONTACTS AND LOCATIONS:
Overall Officials: CAIO VINICIUS G ROMAN TORRES, Principal Investigator — University of Santo Amaro
Locations (1):
- Caio Vinicius Gonçalves Roman Torres, Santos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
the data obtained must be presented in manuscript form to be published in a specialized journal of the area

REFERENCES:
- [Background] Izuora K, Ezeanolue E, Schlauch K, Neubauer M, Gewelber C, Umpierrez G. Impact of periodontal disease on outcomes in diabetes. Contemp Clin Trials. 2015 Mar;41:93-9. doi: 10.1016/j.cct.2015.01.011. Epub 2015 Jan 24. PMID 25623292
- [Result] Simpson TC, Weldon JC, Worthington HV, Needleman I, Wild SH, Moles DR, Stevenson B, Furness S, Iheozor-Ejiofor Z. Treatment of periodontal disease for glycaemic control in people with diabetes mellitus. Cochrane Database Syst Rev. 2015 Nov 6;2015(11):CD004714. doi: 10.1002/14651858.CD004714.pub3. PMID 26545069
- [Result] Wang X, Han X, Guo X, Luo X, Wang D. The effect of periodontal treatment on hemoglobin a1c levels of diabetic patients: a systematic review and meta-analysis. PLoS One. 2014 Sep 25;9(9):e108412. doi: 10.1371/journal.pone.0108412. eCollection 2014. PMID 25255331
- [Result] Pranckeviciene A, Siudikiene J, Ostrauskas R, Machiulskiene V. Long-term effect of periodontal surgery on oral health and metabolic control of diabetics. Clin Oral Investig. 2017 Apr;21(3):735-743. doi: 10.1007/s00784-016-1819-y. Epub 2016 Apr 11. PMID 27068410